CLINICAL TRIAL: NCT03576326
Title: Influence of Financial Incentives on Oral Disease Management in Young Children
Brief Title: BEhavioral EConomics for Oral Health iNnovation Trial
Acronym: BEECON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Los Angeles (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NIDCR 17-084-E UH3DE025514; UH3DE025514 (NIH)
Record Dates: First submitted 2018-05-23; First posted 2018-07-03 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Toothbrushing; Dental Plaque; Parent-Child Relations; Oral Hygiene; Dental Caries
Keywords: Preventive Dentistry; Health Disparities; Health Behavior; Behavioral Economics
MeSH Terms: conditions — Dental Plaque; Dental Caries; Health Behavior

STUDY DESIGN:
Intervention Model Description: Eligible consenting parent-child participant dyads, within strata and permuted blocks, will be randomized in equal allocation to one of two arms. Strata will be based on site and smartphone operating system (iOS or Android).
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent outcomes assessor and PIs will be blinded to participants' group assignment, and participants will be told that the examiner and PIs cannot answer any incentive questions and they should not mention the incentive program to them. (Due to the nature of the intervention, the staff explaining the study arms after randomization and providing the incentive gift cards at follow-up visits cannot be blinded.)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentive Drawing (Experimental): Eligible to earn a weekly drawing entry with different winning probabilities during the 6-month incentive intervention period. Possible winnings depend on toothbrushing performance: low adherence threshold (brushing child's teeth once per day for 7 days in a week) will have an 18% chance of winning $25 and a 1% chance of winning $50 (expected $5 payout); high adherence threshold (brushing twice per day for 14 days in a week) will have a 34% chance of winning $25 and a 3% chance of winning $50 (expected $10 payout).
  Interventions: Behavioral: Drawing Incentive
- Control - Delayed Incentive (No Intervention): No rewards during the first 12 months, but information on toothbrushing performance. After the Month 12 follow-up visit, may opt to participate in a delayed 6-month open label extension to earn the same monetary rewards the intervention group could earn Baseline through Month 6. Not a formal part of this trial, but rather a necessary condition to assure all participating parents/caregivers have the chance to earn the same monetary incentives.

INTERVENTIONS:
Behavioral: Drawing Incentive — The Monetary Reward intervention is a drawing reward, in which participants are eligible for weekly rewards based on toothbrushing performance.
  Arms: Incentive Drawing

SUMMARY:
This Phase II stratified randomized prevention trial will assess the efficacy of a behavioral economic theory-based financial incentive drawing program versus a control regimen to promote early childhood caries (ECC) preventive health behaviors (toothbrushing performance) for young children of predominantly Latino parents/caregivers in Early Head Start (EHS) and day care center programs.

ELIGIBILITY:
Inclusion Criteria:

* Child

  * at least 2 fully erupted teeth
  * enrolled in, or waitlisted for, one of the participating Los Angeles County Early Head Start (EHS) or affiliated day care center or area clinic programs
* Parent/caregiver

  * provide signed and dated informed consent form in English or Spanish
  * agree to comply with all study procedures and be available for the duration of the study
  * aged 18 or older
  * speak either English or Spanish and self-reported ability to read and write either English or Spanish
  * be a parent or caregiver of a child at least 6 months old but less than 4 years (48 months), with at least 2 fully erupted teeth and enrolled in, or waitlisted for, one of the participating Los Angeles County EHS or affiliated day care center or area clinic programs
  * not be planning to move residence for the next 18 months outside the greater Los Angeles area
  * own a smartphone with Google Play or iTunes store app and be willing to download and install the smart powered toothbrush app at the Screening visit and keep it installed for the duration of the project. [If the app cannot be properly installed by the baseline visit, the participant will not be randomized.]
  * be willing to be contacted via text-messaging (SMS) for study related notifications, such as incentives earned or reminders to sync the toothbrush
* Stakeholder

  * be a staff member at a participating study site (e.g. EHS or affiliated day care center)
  * verbally agree to participate after being provided a study information sheet

Exclusion Criteria:

* Child

  * known allergic reaction to components of the study product(s)
  * uncooperative or behaviorally unsuited (assessed during a toothbrush prophylaxis, ASTDD Basic Screening Survey caries screening, and photograph of maxillary incisors at the screening visit)
  * more than 2 crowns on maxillary incisor teeth (teeth# D, E, F, G, or equivalently #52, 51, 61, 62).
  * participated in the BEECON pilot trial
  * a sibling of a child enrolled in the study (the family's oldest child in the eligible age range will be the study child)
  * enrolled in foster care
  * anything else that would place him/her at increased health risk or preclude the individual's full compliance with or completion of the study
* Parent/caregiver

  * participated in the BEECON pilot trial
  * unable or unwilling to install and use the smart powered toothbrush app during the run-in period

Ages: 6 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 244 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Gansky, DrPH, Principal Investigator — University of California, San Francisco; Francisco Ramos-Gomez, DDS, MS, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- Venice Family Clinic Children First Early Head Start, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available.
Supporting Information: Study Protocol
Time Frame: Specifics are undecided but will be in accordance with NIH rules
URL: https://datadryad.org/

REFERENCES:
- [Derived] Ramos-Gomez F, White JS, Lindau HE, Lin TK, Finlayson TL, Liu JX, Gansky SA. Family monetary incentives as a value-based care model for oral hygiene: rationale and design of the BEhavioral EConomics for Oral health iNnovation (BEECON) trial. J Public Health Dent. 2020 Oct 8:10.1111/jphd.12406. doi: 10.1111/jphd.12406. Online ahead of print. PMID 33090505

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Child-Parent Dyads were recruited and Dyad is the unit of analysis Protocol Enrollment number is the number of Dyads recruited, enrolled, and analyzed; total number of participants who Started the study is the number of Individual participants in the study (i.e., 2x number of dyads).
Groups:
- Incentive Drawing: Children; Incentive Drawing: Parents: Eligible to earn a weekly drawing entry with different winning probabilities during the 6-month incentive intervention period. Possible winnings depend on toothbrushing performance: low adherence threshold (brushing child's teeth once per day for 7 days in a week) will have an 18% chance of winning $25 and a 1% chance of winning $50 (expected $5 payout); high adherence threshold (brushing twice per day for 14 days in a week) will have a 34% chance of winning $25 and a 3% chance of winning $50 (expected $10 payout).
  Drawing Incentive: The Monetary Reward intervention is a drawing reward, in which participants are eligible for weekly rewards based on toothbrushing performance.
- Control - Delayed Incentive: Children; Control - Delayed Incentive: Parents: No rewards during the first 12 months, but information on toothbrushing performance. After the Month 12 follow-up visit, may opt to participate in a delayed 6-month open label extension to earn the same monetary rewards the intervention group could earn Baseline through Month 6. Not a formal part of this trial, but rather a necessary condition to assure all participating parents/caregivers have the chance to earn the same monetary incentives.
Period: Overall Study
Arm/Group | Incentive Drawing: Children | Incentive Drawing: Parents | Control - Delayed Incentive: Children | Control - Delayed Incentive: Parents
Started | 122 | 122 | 122 | 122
3 Months | 107 | 107 | 106 | 106
6 Months | 101 | 101 | 103 | 103
Completed | 92 | 92 | 94 | 94
Not Completed | 30 | 30 | 28 | 28

BASELINE CHARACTERISTICS:
Population: Child-Caregiver (Parent) Dyads
Groups:
- Total: Total of all reporting groups
Arm/Group | Incentive Drawing: Children | Incentive Drawing: Parents | Control - Delayed Incentive: Children | Control - Delayed Incentive: Parents | Total
Number analyzed (Participants) | 122 | 122 | 122 | 122 | 488
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 122 | 0 | 122 | 1 | 245
  Between 18 and 65 years | 0 | 122 | 0 | 120 | 242
  >=65 years | 0 | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.6 (0.9) | 32.4 (7.0) | 1.6 (0.8) | 32.7 (6.7) | 17.1 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 117 | 52 | 114 | 346
  Male | 59 | 5 | 70 | 8 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 106 | 106 | 102 | 102 | 416
  Not Hispanic or Latino | 16 | 15 | 20 | 20 | 71
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 4 | 4 | 4 | 4 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 4 | 4 | 6 | 5 | 19
  White | 33 | 34 | 25 | 29 | 121
  More than one race | 3 | 0 | 5 | 0 | 8
  Unknown or Not Reported | 77 | 79 | 82 | 83 | 321
Study Site [Count of Participants; unit: Participants]
  Location A | 26 | 26 | 27 | 27 | 106
  Location B | 87 | 87 | 90 | 90 | 354
  Location C | 9 | 9 | 5 | 5 | 28

OUTCOME MEASURES:

1. Primary Outcome: Toothbrushing Performance
Description: Mean of the number of qualifying half-day episodes per week in which a parent/caregiver brushes a child's teeth. (A Bluetooth-recorded toothbrushing episode qualifies if it lasts at least one minute within one of 14 half-day windows in the week.)
Time Frame: Baseline visit through the Month 6 visit
Population: any post-baseline evaluable data from 0 to 6 months
Measure: Mean (Standard Deviation); unit: qualifying half-day episodes per week
Arm/Group | Control - Delayed Incentive: Parents | Incentive Drawing: Parents
Number analyzed (Participants) | 116 | 116
qualifying half-day episodes per week | 4.6 (2.8) | 5.6 (3.3)

2. Secondary Outcome: Short-term (Immediate) Toothbrushing Performance
Description: Mean number of qualifying half-day episodes per week in which a parent/caregiver brushes a child's teeth.
Time Frame: Baseline visit through the Month 1 visit
Population: any post-baseline evaluable data from 0 to 1 months
Measure: Mean (Standard Deviation); unit: qualifying half-day episodes per week
Arm/Group | Control - Delayed Incentive: Parents | Incentive Drawing: Parents
Number analyzed (Participants) | 111 | 109
qualifying half-day episodes per week | 5.4 (3.2) | 6.2 (3.7)

3. Secondary Outcome: Mid-term Toothbrushing Performance
Description: Mean number of qualifying half-day episodes per week in which a parent/caregiver brushes a child's teeth.
Time Frame: Baseline visit through the Month 3 visit
Population: any post-baseline evaluable data from 0 to 3 months
Measure: Mean (Standard Deviation); unit: qualifying half-day episodes per week
Arm/Group | Control - Delayed Incentive: Parents | Incentive Drawing: Parents
Number analyzed (Participants) | 113 | 112
qualifying half-day episodes per week | 4.9 (3.0) | 5.8 (3.4)

4. Secondary Outcome: Toothbrushing Performance Sustainability
Description: Mean number of qualifying half-day episodes per week in which a parent/caregiver brushes a child's teeth.
Time Frame: Month 6 visit through the Month 12 visit
Population: any post-baseline evaluable data from 6 to 12 months
Measure: Mean (Standard Deviation); unit: qualifying half-day episodes per week
Arm/Group | Control - Delayed Incentive: Parents | Incentive Drawing: Parents
Number analyzed (Participants) | 97 | 98
qualifying half-day episodes per week | 4.3 (2.6) | 4.8 (3.3)

5. Secondary Outcome: Self-efficacy Scale
Description: Caregiver (parent) oral health self-efficacy items (total score ranges 6-30 with higher score indicating more self-efficacy; 6 items each on 1-5 ordinal scale, Albino et al.; Finlayson et al.)
Time Frame: Month 6 visit
Population: some participants did not complete the self-efficacy instrument at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control - Delayed Incentive: Parents | Incentive Drawing: Parents
Number analyzed (Participants) | 103 | 101
score on a scale | 26.4 (2.6) | 25.9 (3.1)

6. Secondary Outcome: Modified Simplified Oral Hygiene Index
Description: Debris Index of the Simplified Oral Hygiene Index for Maxillary Incisors (OHI-MIS) to measure child's plaque on primary maxillary incisor facial (labial) tooth surfaces (mean of 4 ordinal scores each with values ranging from no plaque (1) - which is best - to abundant plaque (4) - which is worst)
Time Frame: Month 6 visit and Month 12 visit
Population: Not all randomized children were available for evaluation at Month 6 and Month 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control - Delayed Incentive: Children | Incentive Drawing: Children
Number analyzed (Participants) | 90 | 86
units on a scale
  Month 6 | 2.2 (0.6) | 2.1 (0.5)
  Month 12: number analyzed (Participants) | 76 | 75
  Month 12 | 2.2 (0.6) | 2.1 (0.6)

7. Secondary Outcome: Change From Baseline in Toothpaste Weight
Description: Change in child's toothpaste pump weight (grams) from each distribution visit (6 months prior). Negative mean values are a decrease from an earlier time to a subsequent time.
Time Frame: From Baseline to Month 6 visit and From Month 6 visit to Month 12 visit
Population: Data were only available for participants who brought toothpaste tube back on follow-up visits at Month 6 and Month 12.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Control - Delayed Incentive: Children | Incentive Drawing: Children
Number analyzed (Participants) | 67 | 66
grams
  Baseline to Month 6 | -44.9 (25.4) | -40.9 (27.7)
  Month 6 to Month 12: number analyzed (Participants) | 43 | 42
  Month 6 to Month 12 | -51.4 (32.5) | -48.0 (32.3)

8. Secondary Outcome: Untreated Caries
Description: Number and percent of children with untreated caries using Association of State and Territorial Dental Directors Basic Screening Survey (ASTDD BSS) binary (yes/no) measure of child's untreated caries status (dt>0)
Time Frame: Month 6 visit and Month 12 visit
Population: Not all randomized children were available for evaluation at Month 6 and Month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Delayed Incentive: Children | Incentive Drawing: Children
Number analyzed (Participants) | 94 | 90
Participants
  Month 6 | 14 | 13
  Month 12: number analyzed (Participants) | 80 | 86
  Month 12 | 9 | 14

9. Secondary Outcome: Caries Experience
Description: Number and percent of children with any history of caries using Association of State and Territorial Dental Directors Basic Screening Survey (ASTDD BSS) binary (yes/no) measure of child's caries experience status (dmft>0)
Time Frame: Month 6 visit and Month 12 visit
Population: Not all randomized children were available for evaluation at Month 6 and Month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Delayed Incentive: Children | Incentive Drawing: Children
Number analyzed (Participants) | 94 | 90
Participants
  Month 6 | 16 | 17
  Month 12: number analyzed (Participants) | 80 | 86
  Month 12 | 12 | 18

10. Secondary Outcome: Severe Caries
Description: Number and percent of children with severe caries experience using Association of State and Territorial Dental Directors Basic Screening Survey (ASTDD BSS) binary (yes/no) measure of child's severe caries experience status (dmft>=4)
Time Frame: Month 6 visit and Month 12 visit
Population: Not all randomized children were available for evaluation at Month 6 and Month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Delayed Incentive: Children | Incentive Drawing: Children
Number analyzed (Participants) | 94 | 90
Participants
  Month 6 | 3 | 5
  Month 12: number analyzed (Participants) | 80 | 86
  Month 12 | 3 | 5

11. Secondary Outcome: Past Year Dental Visit
Description: Number and percent of children with a dental visit in the past 12 months, obtained through Early Head Start ChildPlus database which records child's binary annual dental visit (yes/no) and other required health screenings
Time Frame: Month 12 visit
Population: Data was not systematically recorded in the Early Head Start (EHS) ChildPlus database for individual child participants. EHS reports total number of visits per month but does not record that info for individuals in the EHS ChildPlus database.
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Delayed Incentive: Children | Incentive Drawing: Children
Number analyzed (Participants) | 8 | 6
Participants | 6 | 5

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events were observed for child participants only; parents were not monitored/assessed any of their own adverse events
Arm/Group | Incentive Drawing: Children | Incentive Drawing: Parents | Control - Delayed Incentive: Children | Control - Delayed Incentive: Parents
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/0 | 0/122 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/0 | 0/122 | 0/0
Other Adverse Events (participants affected / at risk) | 3/122 | 0/0 | 5/122 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Incentive Drawing: Children (N=122) | Incentive Drawing: Parents (N=0) | Control - Delayed Incentive: Children (N=122) | Control - Delayed Incentive: Parents (N=0)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 3 (3) | 0 (0) — Fractured/broken tooth due to accident such as falling
Dental infection/abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dental crown (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT03576326/Prot_SAP_000.pdf
  • Informed Consent Form: English (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT03576326/ICF_001.pdf
  • Informed Consent Form: Spanish (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT03576326/ICF_002.pdf